CLINICAL TRIAL: NCT06579118
Title: The Impact of Laughter Yoga on Symptom Management and Quality of Life in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayse Aydin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Tuba Çelik
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Menopause
Keywords: laughter yoga; menopause; symptom; quality of life
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistics expert
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In order to have laughter yoga as a nursing intervention, a "laughter yoga leadership certificate" was obtained by the researcher. Mobile phone numbers were taken to contact the women.Laughter sessions were held in an empty room in the Gynecology outpatient clinic, away from the other rooms indicated by the nurse.A total of 8 sessions of laughter yoga were applied for 4 weeks,2 sessions per week.Before starting laughter yoga, 8 separate WhatsApp groups consisting of approximately 8 people were established to ensure faster and easier communication with women, and information was provided about the sessions and communication was provided. In consultation with the women, the appropriate day, time and program for the session were determined.Sessions will be held twice a week;It was done between 13.00-13.45 on Mondays and Fridays.The sessions were performed in an empty room in the outpatient clinic.A warning sign was hung on the door to avoid being disturbed during the application.
  Interventions: Other: Laughter yoga
- Control group (No Intervention): * Written consent was obtained from pregnant women who agreed to participate in the study.
  * In order to determine the descriptive characteristics of menopausal women, they were asked to fill out the "Personal Information Form", "Menopause Rating Scale" and "Menopause-Specific Quality of Life Scale".
  * After 4 weeks, the process was completed by having women in menopause fill out the "Menopause Symptoms Assessment Scale/MSDS" and "Menopause-Specific Quality of Life Scale/MSDS".

INTERVENTIONS:
Other: Laughter yoga — The women in the experimental group were given laughter yoga sessions by the researcher.
  Arms: Experimental Group

SUMMARY:
This study aimed to assess the impact of laughter yoga intervention on symptomatology and quality of life among postmenopausal women.The research was conducted in a randomized controlled experimental design.

DETAILED DESCRIPTION:
The population of the research consisted of menopausal women who applied to the Gynecology Polyclinic of Atatürk University Health Research and Application Center between 25.08.2023 and 15.12.2023. To determine the sample size of the study, a priori power analysis was performed in the G* Power 3.1.9.7 program. Based on the medium effect size (0.5), the alpha value was determined as 5% and the theoretical power was determined as 95%, and the minimum sample size was determined as 64. The sample of the study consisted of 128 women, 64 experimental and 64 control, who met the research criteria and agreed to participate in the research. However, since 8 people in the experimental group could not continue laughter yoga, the study was completed with 120 women.

Criteria for inclusion in the study

* Entering natural menopause,
* Being over 45 years old,
* Being at least a primary school graduate (in order to be able to fill out the forms),
* Agreeing to participate in the research voluntarily,
* Not having any hearing or vision problems (in order to be able to perform the sessions),
* No diagnosed psychiatric disease,
* Knowing Turkish,
* Having a smart mobile phone
* Being open to communication and cooperation.

Exclusion criteria from the study

• Not continuing with laughter yoga sessions.

Data were collected using the "Personal Information Form," "Menopause Rating Scale," and "Menopause-Specific Quality of Life Scale." Laughter yoga was used as an intervention tool in the research.Participants in the experimental group underwent laughter yoga sessions twice weekly for four weeks, totaling eight sessions.

The data were collected by the researcher through a face-to-face interview in a suitable empty room at Atatürk University Health Research and Application Center Gynecology Polyclinic. In order to enable women to answer the questions comfortably, each woman was interviewed alone in a separate room in the relevant outpatient clinic. Application of the questionnaire and scales took an average of 10-15 minutes for each woman. Before starting the research, women were informed about the purpose, method, rights and responsibilities of the research.

Process steps experimental group

* Written consent was obtained from menopausal women who agreed to participate in the study.
* 10 minutes before starting the laughter yoga, women in menopause were asked to fill out the "Personal Information Form", "Menopause Rating Scale" and "Menopause-Specific Quality of Life Scale" in order to determine their descriptive characteristics.
* A total of 8 sessions of laughter yoga were applied for 4 weeks, 2 sessions per week. The first session lasted 45 minutes, all other sessions lasted an average of 30 minutes. In the first session, laughter yoga, its history, benefits, breathing techniques, laughter yoga exercises were mentioned before the exercises, and in the following sessions, reminders were made and the session ended with laughter yoga exercises and breathing exercises.
* After 4 weeks, the process was completed by having women in menopause fill out the "Menopause Rating Scale" and the "Menopause-Specific Quality of Life Scale".

control group

* Written consent was obtained from pregnant women who agreed to participate in the study.
* In order to determine the descriptive characteristics of menopausal women, they were asked to fill out the "Personal Information Form", "Menopause Symptoms Evaluation Scale" and "Menopause-Specific Quality of Life Scale".
* After 4 weeks, the process was completed by having women in menopause fill out the "Menopause Rating Scale" and "Menopause-Specific Quality of Life Scale".

Data analysis included Skewness and Kurtosis values, frequency and percentage distributions, Chi-square tests, Independent Samples t-test, Paired Samples t-test, Mann-Whitney U test, Wilcoxon signed-rank test, and regression analysis. All ethical principles were adhered to throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Entering natural menopause,
* Being over 45 years old,
* Being at least a primary school graduate (in order to be able to fill out the forms),
* Agreeing to participate in the research voluntarily,
* Not having any hearing or vision problems (in order to be able to perform the sessions),
* No diagnosed psychiatric disease,
* Knowing Turkish,
* Having a smart mobile phone
* Being open to communication and cooperation.

Exclusion Criteria:

* Not continuing with laughter yoga sessions.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Menopause women
Enrollment: 120 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 5 months
  It consists of 10 questions (age, gender, education level, marital status, income status, etc.) prepared by the researcher in line with the literature.
Menopause Rating Scale | 5 months
  The scale, which includes a total of 11 items including menopausal complaints, consists of 3 sub-dimensions. These sub-dimensions are 1-Somatic complaints sub-dimension (items 1,2,3,11), 2-Psychological complaints sub-dimension (items 4,5,6,7), 3-Urogenital complaints sub-dimension (8,9, Article 10). The scale is a 5-point Likert type and each statement is scored as 0: None, 1: Mild, 2: Moderate, 3: Severe and 4: Very severe. The total score of the scale is calculated based on the scores given for each item. The minimum score that can be obtained from the scale is 0, while the maximum score is 44. An increase in the total score obtained from the scale, on the one hand, indicates an increase in the severity of the complaints experienced, and on the other hand, indicates that the quality of life is negatively affected.
Menopause-Specific Quality of Life Scale | 5 months
  It is a Likert type scale containing 29 questions. It consists of four subdomains: vasomotor domain (questions 1-3), psychosocial domain (questions 4-10), physical domain (questions 11-26) and sexual domain (questions 27-29). The complaints that women have experienced in the last month are questioned and the answers to the questions are "yes" or "no". In MÖYÖS, each subdomain score is ranked from 0 to 6. A score of "0" indicates that there are no problems with the issue. A score of "1" indicates that the problem exists and is experienced, but it is not disturbing at all, and scores between "2-6" indicate the severity and increasing degrees of the existing problem. The lowest score that can be obtained from the total of the scale is "0" and the highest score (29X6) is 154. However, evaluation is not made based on the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Aydın, Principal Investigator — Ataturk University
Locations (1):
- Ayşe Aydın, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No